CLINICAL TRIAL: NCT07102485
Title: A Comparison of Labels "Natural Immunity" and "Disease-induced" Immunity
Brief Title: A Comparison of People's Responses to the Labels "Natural Immunity" Versus "Disease-induced Immunity".
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: natimm
Record Dates: First submitted 2025-07-28; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Attitudes
MeSH Terms: conditions — Behavior | interventions — Immunity, Innate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- natural immunity (Placebo Comparator): Label used is standard term "natural immunity"
  Interventions: Other: natural immunity
- disease-induced immunity (Experimental): Label used is "disease-induced immunity"
  Interventions: Other: disease-induced immunity

INTERVENTIONS:
Other: disease-induced immunity — Using a different label for natural immunity, specifically, "disease-induced immunity"
  Arms: disease-induced immunity
Other: natural immunity — Using standard label "natural immunity"
  Arms: natural immunity

SUMMARY:
A comparison of how people respond to the terms "natural immunity" versus "disease-induced immunity".

ELIGIBILITY:
Inclusion Criteria:

* Able to use a computer
* Able to use the internet
* Able to read and respond to questions in English or French
* 18+ years old and living in Canada

Exclusion Criteria:

- not meeting inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2025-07-24 (Estimated); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Opinion about forms of immunity | Immediately after intervention
  Participants indicate their opinion in response to question, "In your opinion, which is better: vaccine-induced immunity or natural/disease-induced immunity?" on a visual analog scale (slider) from 0-100, with 0 = "vaccine-induced immunity is much better," 50 = "both forms of immunity are equally good," 100 = "natural/disease-induced immunity is much better."

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data will be shared on Borealis, Laval University's data repository.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: IPD and supporting information will be available when the report is complete and for an indefinite period of time.
Access Criteria: Anyone with internet access will be able to access public-facing data. Some data may require Borealis registration.
URL: https://borealisdata.ca/